CLINICAL TRIAL: NCT04449380
Title: Randomized, Controlled, Open Label, Phase 2 Clinical Trial of Interferon-β-1a (IFNβ-1a) in COVID-19 Patients
Brief Title: Clinical Study for the Treatment With Interferon-ß-1a (IFNß-1a) of COVID-19 Patients
Acronym: INTERCOP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Futility
Sponsor: Emanuele Bosi (Other)
Responsible Party: Sponsor-Investigator, Emanuele Bosi, Professor, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INTERCOP
Record Dates: First submitted 2020-06-23; First posted 2020-06-26 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: COVID-19 Virus Infection
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This is an interventional, monocentric, phase 2, randomized (2:1), open label, controlled clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IFNβ 1a (Experimental)
  Interventions: Drug: Interferon-ß-1a
- Standard care (Active Comparator)
  Interventions: Combination Product: Standard of Care (SOC)

INTERVENTIONS:
Drug: Interferon-ß-1a — IFNβ-1a will be administered subcutaneously at a dose of 44 mcg (equivalent to 12 million international units), three times per week at least 48 hours apart, for a total of two weeks. All patients will receive a total dose of 264 mcg (72 million international units) under physician control
  Other Names: IFNß-1a
  Arms: IFNβ 1a
Combination Product: Standard of Care (SOC) — Any pharmacological (e.g. antibiotics, etc.) and non-pharmacological (e.g. oxygen, ventilation, etc.) treatments prescribed on clinical grounds
  Other Names: SOC
  Arms: Standard care

SUMMARY:
Pharmacological therapies of proven efficacy in coronavirus disease 2019 (COVID-19) are still lacking.

Since two clinical stages of COVID-19 are emerging, an early one with typical clinical characteristics of a viral infection (fever, malaise, cough) and a later one with pneumonia leading to progressive respiratory failure, associated with heavy, cytokine-mediated, inflammation, an intervention by a compound possessing both antiviral activity and immunomodulatory effects would be most effective at the earliest possible stage.

The purpose of this clinical trial is to test the efficacy of Interferon-β-1a (IFNβ-1a), in COVID-19 patients in an open label, randomized clinical trial.

The design of the study is to test IFNβ-1a in addition to standard of care compared with standard of care alone.

The primary outcome is the time to negative conversion of Severe Acute Respiratory Syndrome-CoronaVirus-2 (SARS-CoV-2) nasopharyngeal swabs.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent signed
2. Patients hospitalized with confirmed swab RT-PCR detection of SARS-CoV-2
3. X-ray and/or CT diagnosed pneumonia
4. Age >=18 years
5. Clinical status defined as 3, 4 or 5 on the 7-point ordinal scale

Exclusion Criteria:

1. Known allergy or hypersensitivity to IFNß-1a or IFNß-1b
2. Presence of severe concomitant illnesses/medical conditions that in the physician opinion do not allow participation to the study
3. Pregnant or lactating females
4. History of major depression disorder or suicidal attempt or suicidal ideation
5. Spontaneous blood alanine aminotransferase/aspartate aminotransferase (ALT/AST) levels > 5 times the upper limit of normal
6. Clinical status defined as 1, 2, or 6 on the 7-point ordinal scale

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Time to negative conversion of SARS-CoV-2 nasopharyngeal swab | From baseline to day 29
  Viral load will be measured by Real Time-Polymerase Chain Reaction (RT-PCR)

SECONDARY OUTCOMES:
Improvement in clinical severity score (a) | Baseline, days 7, 15, 21, 29
  Defined as percentage of patients reporting each severity rating on a 7-point ordinal scale
Improvement in clinical severity score (b) | Baseline, days 7, 15, 21, 29
  Defined as the time to clinical improvement of two points from the time of randomization on a 7-category ordinal scale or live discharge from the hospital, whichever comes first
Incidence of new oxygen use, non-invasive ventilation, or high flow oxygen devices during the trial | From baseline to day 29
Oxygenation free days in the first 28 days | From baseline to day 29
Ventilator free days in the first 28 days | From baseline to day 29
Incidence of new mechanical ventilation use during the trial | From baseline to day 29
Number of patients transferred to Intensive Care Unit (ICU) | From baseline to day 29
Mortality rate | From baseline to day 29
Changes from baseline in pulmonary computed tomography (CT) imaging severity score | Baseline, day 21; extra follow up at 90 days
  Measured with artificial intelligence and expressed as cc and percent values of diseased lung (lung consolidation, ground glass opacities and disease free)
Duration of hospital stay expressed in days | From baseline to day 29
Viral load measured on plasma with RT-PCR | Baseline, days 3, 5, 7, 9, 11, 13, 15, 21, 29

OTHER OUTCOMES:
Plasma and peripheral blood mononuclear cell messenger-RNA (mRNA) expression profile of interferon stimulated genes (ISG) | Baseline, day 15
Antibodies to SARS-CoV-2 | Baseline, days 7, 15, 29
Antibodies to IFN-β1a | Baseline, days 7, 15, 29

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele Bosi, Professor, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

REFERENCES:
- [Derived] Bosi E, Bosi C, Rovere Querini P, Mancini N, Calori G, Ruggeri A, Canzonieri C, Callegaro L, Clementi M, De Cobelli F, Filippi M, Bregni M. Interferon beta-1a (IFNbeta-1a) in COVID-19 patients (INTERCOP): study protocol for a randomized controlled trial. Trials. 2020 Nov 23;21(1):939. doi: 10.1186/s13063-020-04864-4. PMID 33225960